CLINICAL TRIAL: NCT05234476
Title: A Randomized Controlled Trial of Behavioral Activation Plus Savoring for University Students With Positive Valence Dysregulation
Brief Title: Behavioral Activation Plus Savoring for University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Methodist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-118
Record Dates: First submitted 2021-10-08; First posted 2022-02-10 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Mood; Anhedonia; Depression
MeSH Terms: conditions — Anhedonia; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation plus Savoring (Experimental): Individuals in this intervention will complete two sessions of behavioral activation, where they will be provided psychoeducation on behavioral models of mood, schedule activities, and discuss barriers to completion. Additionally, they will practice savoring as a cognitive strategy to increase positive emotions with a study therapist.
  Interventions: Behavioral: Behavioral Activation plus Savoring
- Empathic Listening (Active Comparator): Individuals in the active control condition will complete two sessions of reflecting on tracking their mood and empathic listening with a study therapist.
  Interventions: Behavioral: Empathic Listening

INTERVENTIONS:
Behavioral: Behavioral Activation plus Savoring — Individuals in this intervention will complete two sessions of behavioral activation, where they will be provided psychoeducation on behavioral models of mood, schedule activities, and discuss barriers to completion. Additionally, they will practice savoring as a cognitive strategy to increase positive emotions with a study therapist.
  Arms: Behavioral Activation plus Savoring
Behavioral: Empathic Listening — Individuals in the active control condition will complete two sessions of reflecting on tracking their mood and empathic listening with a study therapist.
  Arms: Empathic Listening

SUMMARY:
The current investigation aims to examine whether a brief, two-session, virtual behavioral activation plus savoring intervention will increase daily positive emotion in university students.

DETAILED DESCRIPTION:
Experiences of positive emotions are often unchanged following standard psychotherapy. To address this, the current investigation aims to enhance traditional brief behavioral activation with savoring, an emotion regulation strategy specifically targeting positive emotion, or affect, for university students endorsing low levels of the symptom. Individuals will be randomized to either a two-session behavioral activation plus savoring intervention or two sessions of empathic listening. Daily levels of positive emotions will be assessed throughout the study and for one week prior to and completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* University student
* Own a smartphone
* Positive affect score less than 32 on the Positive and Negative Affect Schedule, Short Form (PANAS-SF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Positive Emotions: Modified Differential Emotions Scale (mDES; Fredrickson et al., 2003) | Change from first session to post-treatment (14 days)
  Positive mood, as measured by the mDES, will be collected two times a day. Participants will be asked to rate their level of positive mood in the moment. Positive mood will be collected on a daily basis throughout the study and change in reported positive emotions will be assessed.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | Change from baseline to post-treatment (21 days)
  Change in reported symptoms of positive and negative affect following the intervention
Depression, Anxiety, and Stress Scale (DASS-21) | Change from baseline to post-treatment (21 days)
  Change in self-reported symptoms of depression, anxiety, and stress following the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kumar D, Corner S, Kim R, Meuret A. A randomized controlled trial of brief behavioral activation plus savoring for positive affect dysregulation in university students. Behav Res Ther. 2024 Jun;177:104525. doi: 10.1016/j.brat.2024.104525. Epub 2024 Mar 24. PMID 38653177